CLINICAL TRIAL: NCT00739544
Title: Examination of Healthy Female Subjects in the Project: Disposing Factors for Chronic Pain After Operation for Breast Cancer
Brief Title: Chronic Pain After Operation for Breast Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Breast Cancer Cooperative Group (Other); Danish Cancer Society (Other)
Responsible Party: Rune Gärtner MD, Department of Breast Cancer Surgery, RH, Copenhagen University, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: RH2101project.1.2008
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Pain Threshold
Keywords: Reference Values; Sensory Thresholds; Pain Threshold; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Quantitative sensory testing (QST) of healthy women to create reference values for QST evaluation of women treated for breast cancer
  Interventions: Other: 1

INTERVENTIONS:
Other: 1 — Testing with thermal sensor testing device, von Frey filaments, cotton wisp, turning fork, pressure gauge device

SUMMARY:
The purpose of this study is to identify intraindividual as well as iatrogenic factors disposing for the development of chronic and acute pains after surgery for breast cancer in order to improve treatment and prevent the development of acute and chronic postoperative pains.

DETAILED DESCRIPTION:
Surgery for breast cancer is followed by acute undesirable sequelae (pain, nausea, vomiting, psycho-social adaptation) and late sequelae with discomfort or more severe neuropathic pain problems in the surgical area due to nerve damage or adjuvant-/radiotherapy. The late sequelae occur in 30-50% of patients but the exact mechanisms (preoperative disposing factors, intraoperative nerve damage/inflammatory response), acute postoperative pain and psychosocial factors remain to be determined in large, detailed, well-described studies, including stratification to modern breast cancer treatment (sentinel node strategy/ radiotherapy/ chemotherapy). The present study will describe in detail preoperative psychosocial/genetic pain mechanisms, intraoperative technique, multi-modal anaesthesia and opioid-reduced analgesia with a detailed, early and late postoperative follow-up with neurophysiological assessment in the surgical area and randomised studies on preventive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women

Exclusion Criteria:

* Pregnancy
* Lactating

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Reference values on: Cold and cold detection threshold,Paradoxical heat sensation,Thermal sensory limen procedure,Cold and heat pain threshold,Mechanical detection and pain threshold and sensitivity,Vibration detection threshold,Pressure pain threshold | From 08-20-2008 to 11-1-2008 test is performed two times with app one week in between

CONTACTS AND LOCATIONS:
Overall Officials: Niels Kroman, MD, DMSc, Study Director — Department of Breast Surgery, Centre of Head and Orthopaedics, Rigshospitalet (University of Copenhagen), Denmark; Henrik Kehlet, MD Ph.D DMSc, Study Chair — Section for Surgical Pathophysiology, Juliane Marie Centre, Rigshospitalet (University of Copenhagen), Denmark
Locations (1):
- Department of Breast Surgery, Centre of Head and Orthopaedics, Rigshospitalet (university of Copenhagen), Copenhagen, Denmark